CLINICAL TRIAL: NCT07279285
Title: The Effect of a Sugar-free-flavored-sweet-tasting-solution on Pain Associated With Dental Injections in Pediatric Patients
Brief Title: Sweet-Tasting Solution Versus Placebo to Reduce Pain During Local Anesthetic Injection in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Lamis D. Rajab, Prof, University of Jordan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UJordanLamis
Record Dates: First submitted 2025-11-18; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Injection Pain; Local Anesthesia Infiltration; Pain; Injection Pain Prevention; Pediatric Patients
Keywords: clinical trial; sugar-free solution; local anesthesia pain; dental pain; injection pain; children dental pain; split-mouth; sugar-free flavored sweet tasting solution; SFSS; dental fear reduction; dental fear; dental anxiety
MeSH Terms: conditions — Pain; Toothache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugar-free-flavored sweet tasting solution Group (Active Comparator)
  Interventions: Other: Sugar-free-flavored sweet tasting solution
- Placebo Group (Placebo Comparator)
  Interventions: Other: Placebo (sterile-water)

INTERVENTIONS:
Other: Sugar-free-flavored sweet tasting solution — A sugar-free-flavored sweet tasting solution that is anticipated to reduce the pain of local anaesthesia injections
  Arms: Sugar-free-flavored sweet tasting solution Group
Other: Placebo (sterile-water) — Placebo (sterile water)
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to learn whether applying a sugar-free flavored sweet solution (SFSS) before local anesthesia helps reduce injection pain in children.

The main question it aims to answer is:

Does SFSS reduce pain during dental local anesthesia compared to a placebo (plain water)? Researchers will compare the use of SFSS and a placebo to see which results in lower pain scores.

Participants will:

Receive SFSS or placebo before local anesthesia during two dental visits Have their pain measured using self-reported and observational pain scales Have their heart rate monitored during the procedure

ELIGIBILITY:
Inclusion Criteria:

1. Children who are 6-12 years of age.
2. Children classified as ASA1 according to the American Society of Anesthesiologists.
3. Children who have positive (Class III) or definitely positive (Class IV) behavior during preoperative behavioral assessments according to the Frankl Scale.
4. Children who required bilateral local anesthesia infiltration injections on primary or permanent teeth either in the maxilla or mandible for dental treatment (different types of restoration, stainless steel crowns, pulp therapy, and extractions).
5. Children with positive consent forms (signed and approved by their parents/ legal guardians) and attended the appointment.

Exclusion Criteria:

1. Children who had a history of unpleasant experiences in dental settings.
2. Children who had a history of unpleasant experience with local anesthesia injection.
3. The presence of medically or developmentally compromising conditions.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported pain using faces pain scale-revised (FPS-r) | Immediately after local anesthetic injection
  Pain intensity measured using the Faces Pain Scale - Revised (FPS-R), ranging from 0 to 10, where higher scores indicate greater pain.
Observer-reported pain using Revised Face, Legs, Activity, Cry, Consolability Scale | During administration of the local anesthetic injection
  Pain behavior measured using the Face, Legs, Activity, Cry, Consolability - Revised (FLACC-R) Scale, scored from 0 to 10, where higher scores indicate greater pain-related distress.
Physiological-Heart Rate | Baseline and During Injection
  Changes in heart rate measured in beats per minute (bpm); increases in heart rate indicate higher physiological arousal associated with pain

IPD SHARING:
Plan to Share IPD: Yes